CLINICAL TRIAL: NCT00171353
Title: A Study to Describe Vascular and Renal Effects and Safety of Valsartan 80 and 160 mg in Arterial Hypertension Patients
Brief Title: A Study to Describe Vascular and Renal Effects and Safety of Valsartan in Patients With High Blood Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVAL489ARU01
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Hypertension
Keywords: arterial hypertension; albuminuria; valsartan
MeSH Terms: conditions — Hypertension; Albuminuria | interventions — Valsartan

INTERVENTIONS:
Drug: valsartan

SUMMARY:
One hundred twenty patients with arterial hypertension and albuminuria (some amount of albumin in urine) are given valsartan 80 mg and then160 mg to normalize blood pressure. Hydrochlorothiazide (diuretic) 12.5-25 mg added if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Arterial hypertension without previous regular treatment
* Urinary albumin excretion rate above 30 mg / 24h
* 30-65 years old

Exclusion Criteria:

* Reno-vascular arterial hypertension
* Therapy resistant edema
* Chronic heart failure, angina pectoris
* Diabetes mellitus

Other protocol-defined exclusion criteria may apply

Ages: 30 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2004-07; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in urine albumin excretion after 24 weeks
Change from baseline in an ultrasound measurement of blood flow after 24 weeks

SECONDARY OUTCOMES:
Effect of blood pressure changes on urine albumin excretion rate and blood vessel function

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, Basel, Switzerland